CLINICAL TRIAL: NCT03488992
Title: Effect of a Multivitamin/Multimineral/Phytochemical Dietary Supplement on Indices of Human Health
Brief Title: Effect of a MVM Dietary Supplement on Indices of Human Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USANA Health Sciences (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16MHHU
Record Dates: First submitted 2017-03-02; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Metabolic Syndrome
Keywords: dietary supplement, cardiovascular health, oxidative stress
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MVM/phytochemical supplement (Experimental): a multi-vitamin, multi-mineral, phytochemical supplement
  Interventions: Dietary Supplement: MVM/phytochemical supplement
- Placebo (Placebo Comparator): a placebo tablet (microcrystalline cellulose) identical in size, shape and color to the treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: MVM/phytochemical supplement — Consumption of an MVM/phytochemical supplement for 8 weeks
  Arms: MVM/phytochemical supplement
Dietary Supplement: Placebo — Consumption of a placebo tablet identical in size, shape and color to the treatment tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the health benefits of a recently developed multimineral/multivitamin/phytochemical (MVM/phytochemical) nutritional supplement. This newly developed supplement - an advancement of a previous formula designed to enhance human health by providing RDA-levels of essential vitamins and minerals - contains eight phytochemicals selected to address fruit and vegetable undernutrition, and chosen on the basis that: 1) published research from cell culture, animal model and, when available, human clinical work, suggests that it may benefit human health, and 2) it is considered safe for human ingestion at proposed levels of consumption.

DETAILED DESCRIPTION:
This study will be an eight-week, randomized, placebo controlled, parallel arm clinical trial to compare markers of nutritional, inflammatory and oxidative status, cardiovascular and neurological health as well as microbial status in subjects consuming a novel multivitamin/multimineral/phytochemical (MVM/phytochemical) supplement compared to subjects consuming a placebo tablet. In addition, this study will evaluate whether the MVM/phytochemical supplement improves subjects sense of well-being as evaluated by a quality-of-life survey. The study will aim to enroll 112 consenting men and women characterized as having metabolic syndrome. Potential subjects will be recruited through flyers, newspapers and advertisements placed throughout the community. Consented subjects will undergo a 28-day washout, followed by a 56-day trial period. Biological samples (blood, urine, stool, saliva) will be collected at baseline (day 0) and at day 56. Diet and exercise history, as well as a quality of life survey, will be collected at these time points as well. Risk to participants is expected to be minimal and will be outlined through an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 29.9 to 40 kg/m2 ±1 kg/m2
* Waist measurement for males ≥ 102 cm (40 inches) or for females ≥ 89 cm (35 inches)
* two or more of the following risk factors:

  * Elevated blood pressure ( 130/85 mm Hg)
  * Fasting elevated triglycerides > 1.69 mmol/L ( 150 mg/dL)
  * Elevated fasting glucose > 5.56 mmol/L ( 100 mg/dL) and <7.0 mmol/L (<126 mg/dL)
  * Low HDL cholesterol <1.29 mmol/L ( 50 mg/dL) for females, and <1.03 mmol/L ( 40 mg/dL) for males
* Not currently taking a multivitamin/mineral, antioxidant supplement, or other dietary supplements or are willing to wash out for 4 weeks before enrollment

Exclusion Criteria:

* Pregnant and/ or lactating females or females trying to become pregnant
* Use of lipid lowering medications
* Lipid lowering OTC or herbal supplements within 3 weeks of enrollment
* Use of conventional multivitamin/mineral, antioxidant supplements or other dietary supplements within four weeks prior to enrollment
* Insulin-dependent Type I and Type II diabetics
* Diabetic men > 45 years and diabetic women > 55 years
* Metformin or other diabetes medications are prohibited in this study
* Type II diabetes controlled by diet and/or exercise
* Elevated blood pressure ( 160/95 mm Hg) at screening
* Individuals with a history of coronary artery disease, previous myocardial infarction, peripheral vascular disease, or atherosclerosis
* Men above 50 years and women above 60 years who have a 10-year risk of cardiovascular event FRS between 10% and 19% (inclusive) at screening and who present with one of the following LDL-C > 3.5 mmol/L, TC/HDL-C ratio > 5.0, or hs-CRP > 2 mg/L
* Individuals with a 10-year risk of cardiovascular event FRS < 10% at screening and present with LDL-C > 5.0 mmol/L or TC/HDL-C ratio > 6.0
* Participants taking blood thinners
* Participants with stomach ulcers, gall stones, or bile duct obstruction

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
HDL Cholesterol | 8 weeks
  Effect of MVM/Phytochemical Supplement on HDL-cholesterol levels compared to placebo

SECONDARY OUTCOMES:
Inflammation | 8 weeks
  change in inflammatory markers between MVM/Phytochemical Supplement and placebo including circulating levels of IL-1b, TNF-a, and IFNg
Oxidative Stress | 8 weeks
  change in oxidative stress markers between MVM/Phytochemical Supplement and placebo including antioxidant enzyme activity (SOD, Catalase, GSH-Px) and markers of oxidative stress (GSH/GSSG, 8-isoprostanes)
Cardiovascular Health | 8 weeks
  change in markers of cardiovascular health between MVM/Phytochemical including Cholesterol levels Supplement and placebo (LDL, HDL, total cholesterol, homocysteine)
Nutritional status | 8 weeks
  change in markers of nutritional status between MVM/Phytochemical Supplement and placebo including vitamins A,D,E,K,C,B6,B12 and folate)
Neurological Health | 8 weeks
  change in markers of neurological health between MVM/Phytochemical Supplement and placebo
Microbiome | 8 weeks
  change in microbiome between MVM/Phytochemical Supplement and placebo using 16s analysis
Quality of Life | 8 weeks
  difference in self-perceived quality of life between MVM/Phytochemical Supplement and placebo using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mark Levy, Principal Investigator — USANA Health Sciences
Locations (1):
- KGK Synergize, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No